CLINICAL TRIAL: NCT05028400
Title: Intraoperative Laser Speckle Contrast Imaging to Assess Blood Flow During Neurosurgery
Acronym: LSCI-NSURG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LSCI-NSURG
Record Dates: First submitted 2021-08-24; First posted 2021-08-31 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Aneurysm; AVM; Dural Arteriovenous Fistula; Glioma; Meningioma; Metastasis
MeSH Terms: conditions — Aneurysm; Central Nervous System Vascular Malformations; Glioma; Meningioma; Neoplasm Metastasis | interventions — Laser Speckle Contrast Imaging

STUDY DESIGN:
Intervention Model Description: Laser speckle contrast imaging (LSCI)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Laser speckle contrast imaging (LSCI) (Experimental): LSCI videos will be recorded automatically intraoperatively in each patient before, during, and after ICGA and/or FA in the same surgical field of view to guarantee comparability of the methods.
  Interventions: Device: Laser speckle contrast imaging (LSCI)

INTERVENTIONS:
Device: Laser speckle contrast imaging (LSCI) — LSCI videos will be recorded automatically intraoperatively in each patient before, during, and after ICGA and/or FA in the same surgical field of view to guarantee comparability of the methods.

SUMMARY:
Cerebral blood flow (CBF) is of paramount importance to human brain function, as the brain relies on a continuous blood supply to meet its energy needs. Blockage of a cerebral blood vessel during neurosurgery, even if transient and short-lived, may result in irreversible brain tissue damage (i.e. stroke) and loss of cortical function, if not identified quickly enough.

Laser speckle contrast imaging (LSCI) has been demonstrated to provide the ability to visualize flow in vessels in real time and continuously without the need for contrast agents. In LSCI, the tissue of interest is illuminated with low power laser light at red or near infrared wavelengths and the light reflected from the tissue surface is imaged onto a camera. The resulting images are laser speckle patterns and a computer processes the images to produce speckle contrast images, which are images of the motion within the field of view (ie, blood flow).

The purpose of this clinical investigation is to assess the usefulness and accuracy of LSCI compared to ICGA and/or FA during neurovascular surgery. LSCI videos will be recorded automatically intraoperatively in each patient before, during, and after ICGA and/or FA in the same surgical field of view to guarantee comparability of the methods.

DETAILED DESCRIPTION:
Cerebral blood flow (CBF) is of paramount importance to human brain function, as the brain relies on a continuous blood supply to meet its energy needs. Blockage of a cerebral blood vessel during neurosurgery, even if transient and short-lived, may result in irreversible brain tissue damage (i.e. stroke) and loss of cortical function, if not identified quickly enough.

Neurosurgery involves the treatment of blood-vessel related pathologies within the brain, like intracranial aneurysms, arteriovenous malformations and dural arteriovenous fistulas, but also the handling of vessels during brain tumor resections. For these operations, assessment of flow in vessels is of paramount importance. So far, the surgeon can not "see" blood flowing inside the artery or vein. Real-time flow visualization during surgery could help neurosurgeons better understand the consequences of vascular occlusion events during surgery, recognize potential adverse complications, and thus prompt timely intervention to reduce the risk of stroke. The current standard for visualizing flow in arteries during surgery is indocyanine green angiography (ICGA) and fluorescein angiography (FA), which involves administering a bolus of fluorescent dye intravenously and imaging the wash-in of the dye to determine which vessels are perfused. Both ICGA and FA provide only a punctual view of perfusion over several seconds, being far away from a continuous assessment.

Laser speckle contrast imaging (LSCI) has been demonstrated to provide the ability to visualize flow in vessels in real time and continuously without the need for contrast agents. In LSCI, the tissue of interest is illuminated with low power laser light at red or near infrared wavelengths and the light reflected from the tissue surface is imaged onto a camera. The resulting images are laser speckle patterns and a computer processes the images to produce speckle contrast images, which are images of the motion within the field of view (ie, blood flow).

With these properties LSCI has the potential to deliver for the first time continuous visualisation of blood flow in large and small vessels and to overcome limitations of ICGA and FA. LSCI is an established technique for studies of CBF and has predominantly been used to study microcirculation of the cerebral cortex during neurosurgical procedures. However, the spatial resolution in the clinical setting and its accuracy compared to ICGA and FA are unclear.

The purpose of this clinical investigation is to assess the usefulness and accuracy of LSCI compared to ICGA and/or FA during neurovascular surgery. LSCI videos will be recorded automatically intraoperatively in each patient before, during, and after ICGA and/or FA in the same surgical field of view to guarantee comparability of the methods.

ELIGIBILITY:
Inclusion Criteria:

* Vascular pathology of the brain or brain tumors requiring elective microsurgical treatment (e.g., aneurysm, arteriovenous malformation, dural arteriovenous fistula, glioma, meningioma, metastasis)
* Adults (18 years or older)
* Informed consent signed by the subject

Exclusion Criteria:

• Patients lacking capacity to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-03-11 (Actual); Study Completion 2022-03-11 (Actual)

PRIMARY OUTCOMES:
Agreement of ICG/FA and LSCI-findings | During surgery
  Agreement of ICG/FA and LSCI-findings determinating flow in exposed vessels classified as no flow, delayed flow, normal flow

SECONDARY OUTCOMES:
Vessels examined with Laser speckle contrast imaging (LSCI) | During surgery
  Vessels examined with Laser speckle contrast imaging (LSCI)
Vessels examined with Indocyanine green angiography (ICGA) | During surgery
  Vessels examined with Indocyanine green angiography (ICGA)
Vessels examined with Fluorescein angiography (FA) | During surgery
  Vessels examined with Fluorescein angiography

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Raabe, MD, Principal Investigator — Study Principal Investigator
Locations (1):
- Department of Neurosurgery, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No